CLINICAL TRIAL: NCT05674773
Title: Endoscopic and Surgical Treatment Outcomes of Colitis-associated Advanced Neoplasia: a Multicenter Cohort Study
Brief Title: Treatment Outcomes of Advanced Neoplasia in IBD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other); Jeroen Bosch Ziekenhuis (Other); University Medical Center Groningen (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam UMC, location VUmc (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-3219
Record Dates: First submitted 2022-12-19; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD patients with advanced neoplasia: IBD patients with advanced neoplasia (high-grade dysplasia or colorectal cancer) treated with:
  * proctocolectomy
  * (sub)total colectomy
  * partial colectomy
  * endoscopic resection
  Interventions: Procedure: Endoscopic or surgical resection

INTERVENTIONS:
Procedure: Endoscopic or surgical resection — endoscopic or surgical (partial, (sub)total, proctocolectomy) resection

SUMMARY:
In this study, we aimed to (1) compare cumulative incidences of synchronous and metachronous colorectal neoplasia as well as mortality following AN in CD and UC patients who underwent proctocolectomy, (sub)total colectomy, partial colectomy or endoscopic resection, and (2) to determine factors associated with AN treatment choice.

DETAILED DESCRIPTION:
In this retrospective multicenter cohort study, using PALGA (the Dutch nationwide pathology databank), partial colectomy yielded a similar metachronous neoplasia risk compared to (sub)total colectomy after treatment of advanced neoplasia in inflammatory bowel disease. High metachronous neoplasia rates after endoscopic resection underline the importance of strict subsequent endoscopic surveillance.

ELIGIBILITY:
Inclusion Criteria:

* IBD (ulcerative colitis (UC), CD or IBD-unclassified (IBD-U))
* Histological diagnosis of colorectal AN
* Available treatment data

Exclusion Criteria:

* Familial CRC syndrome
* AN prior to IBD diagnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: IBD patients with advanced neoplasia
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Synchronous | up to 6 months
  defined as co-existence of two or more neoplastic colorectal lesions detected in the initial resection specimen or up to 6 months after treatment of the index lesion, categorized in (a) any neoplasia (independent of grade) and (b) only AN
Metachronous (advanced) neoplasia | up to 30 years
  defined as colorectal neoplasia detected >6 months after treatment of index AN, categorized in (a) any neoplasia (independent of grade) and (b) only AN, including the impact of IBD type

SECONDARY OUTCOMES:
All-cause mortality | up to 30 years
  All-cause mortality
Associations with treatment choice | up to 30 years
  Clinical and disease characteristics associated with AN treatment choice

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hoentjen, MD, PhD, Principal Investigator — Radboudumc and University of Alberta
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data available upon reasonable request.